CLINICAL TRIAL: NCT07248111
Title: Effectiveness of the Mindful Compassion Care Program for Healthcare Professionals in Oncology and Palliative Care: a Randomized Controlled Trial With a Qualitative Component
Brief Title: Effectiveness of the Mindful Compassion Care Program for Healthcare Professionals in Oncology and Palliative Care
Acronym: MCCP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Collaborators: St. John's University, Rome, Italy (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 390/2025/SPER/IRCCS
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-09

CONDITIONS: Professional Quality of Life; Palliative Care; Oncology
Keywords: mindfulness; self-compassion; emotional regulation; supportive care; mental health promotion
MeSH Terms: conditions — Neoplasms; Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindful Compassion Care Program (MCCP) (Experimental)
  Interventions: Behavioral: MCCP
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: MCCP — The MCCP is a structured seven-week group intervention integrating elements from Mindfulness-Based Cognitive Therapy (MBCT), Mindfulness-Based Stress Reduction (MBSR), and Compassion-Focused Therapy (CFT). The program consists of six 90-minute weekly sessions plus one intensive 4.5-hour session. Sessions include mindfulness meditation, breathing exercises, yoga practices, imagery techniques, and compassion-focused activities. Daily home practice is supported through guided audio tracks and worksheets. The intervention is delivered in small groups (up to 15 participants) by psychotherapists specifically trained for the MCCP as part of the study.
  Arms: Mindful Compassion Care Program (MCCP)

SUMMARY:
This randomized controlled trial aims to evaluate the effectiveness of the Mindful Compassion Care Program (MCCP), a mindfulness- and compassion-based intervention designed to enhance the emotional and professional well-being of healthcare professionals (HPs). The study adopts a multi-center, open-label, randomized, parallel-group, superiority design and includes HPs (physicians, nurses, and nursing assistants) involved in the clinical care of cancer patients across different settings and disease phases. Eligible participants must not have attended MBSR or other mindfulness-/compassion-based interventions in the preceding six months.

The RCT has a primary objective of assessing the MCCP's effectiveness in increasing positive emotions and reducing negative emotions among HPs working in oncology and palliative care. Secondary objectives include evaluating improvements in professional quality of life and self-compassion. After providing informed consent, HPs will be randomized to receive either the MCCP (experimental group) or no intervention (control group).

DETAILED DESCRIPTION:
The study includes an embedded qualitative component designed to explore the acceptability and perceived value of the MCCP from the perspective of healthcare professionals who received the intervention. Qualitative data will be collected through focus groups conducted with a purposive sub-sample of RCT participants. Participation in the focus groups will be voluntary. This purposive sampling strategy is appropriate as it allows the inclusion of individuals capable of providing rich, relevant, and diverse insights into their experiences with the MCCP and its perceived impact.

ELIGIBILITY:
Inclusion Criteria:

* Being a healthcare professional (physicians, nurses, or nursing assistants) involved in the clinical management of cancer patients across different care settings and illness phases.
* Age ≥ 18 years

Exclusion Criteria:

* HPs must not have attended MBSR or other mindfulness/compassion-based interventions, including in educational or clinical settings, involving activities similar to those in the present study in the previous six months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in affectivity (Positive and Negative Affect Schedule, PANAS composite score: Positive - Negative) | baseline, 8 weeks
  The PANAS is a 20-item self-reported questionnaire assessing positive and negative emotions. The composite score (Positive - Negative) will be calculated for each participant. Positive affectivity refers to emotions such as joy or contentment, whereas negative affectivity refers to emotions such as anger, fear, or sadness. Higher scores indicate greater positive affectivity.

SECONDARY OUTCOMES:
Improvement in Professional Quality of Life | baseline, 8 weeks, 6 month
  Measured using the Professional Quality of Life Scale (ProQOL, Version 5), a 30-item self-reported questionnaire. It assesses three subscales: Compassion Satisfaction (CS), Burnout, and Secondary Traumatic Stress (STS). Higher CS scores indicate improved professional well-being, while lower Burnout and STS scores indicate reduced professional fatigue and stress. The change in scores from T0 to T1 and T2 will quantify improvement.
Improvement in Self-Compassion | baseline, 8 weeks, 6 month
  Measured using the Self-Compassion Scale (SCS), a 26-item self-administered questionnaire covering six components: Self-Kindness, Self-Judgment, Common Humanity, Isolation, Mindfulness, and Over-Identification. The total score is the mean of the six subscales (range 1-5), with higher scores indicating greater self-compassion. The change in scores from T0 to T1 and T2 will indicate the degree of improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Loredana Buonaccorso, MD, Principal Investigator — Azienda USL - IRCCS di Reggio Emilia
Locations (1):
- Azienda USL IRCCS di Reggio Emilia, Reggio Emilia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Orellana-Rios CL, Radbruch L, Kern M, Regel YU, Anton A, Sinclair S, Schmidt S. Mindfulness and compassion-oriented practices at work reduce distress and enhance self-care of palliative care teams: a mixed-method evaluation of an "on the job" program. BMC Palliat Care. 2017 Jul 6;17(1):3. doi: 10.1186/s12904-017-0219-7. PMID 28683799
- [Background] Watts KJ, O'Connor M, Johnson CE, Breen LJ, Kane RT, Choules K, Doyle C, Buchanan G, Yuen K. Mindfulness-Based Compassion Training for Health Professionals Providing End-of-Life Care: Impact, Feasibility, and Acceptability. J Palliat Med. 2021 Sep;24(9):1364-1374. doi: 10.1089/jpm.2020.0358. Epub 2021 Mar 5. PMID 33666500
- [Background] Kamal AH, Bull JH, Wolf SP, Swetz KM, Shanafelt TD, Ast K, Kavalieratos D, Sinclair CT. Prevalence and Predictors of Burnout Among Hospice and Palliative Care Clinicians in the U.S. J Pain Symptom Manage. 2020 May;59(5):e6-e13. doi: 10.1016/j.jpainsymman.2019.11.017. Epub 2019 Nov 26. PMID 31778784
- [Background] Hlubocky FJ, Taylor LP, Marron JM, Spence RA, McGinnis MM, Brown RF, McFarland DC, Tetzlaff ED, Gallagher CM, Rosenberg AR, Popp B, Dragnev K, Bosserman LD, Dudzinski DM, Smith S, Chatwal M, Patel MI, Markham MJ, Levit K, Bruera E, Epstein RM, Brown M, Back AL, Shanafelt TD, Kamal AH. A Call to Action: Ethics Committee Roundtable Recommendations for Addressing Burnout and Moral Distress in Oncology. JCO Oncol Pract. 2020 Apr;16(4):191-199. doi: 10.1200/JOP.19.00806. Epub 2020 Mar 30. PMID 32223701
- [Background] Ho AHY, Tan-Ho G, Ngo TA, Ong G, Chong PH, Dignadice D, Potash J. A Novel Mindful-Compassion Art-Based Therapy for Reducing Burnout and Promoting Resilience Among Healthcare Workers: Findings From a Waitlist Randomized Control Trial. Front Psychol. 2021 Oct 21;12:744443. doi: 10.3389/fpsyg.2021.744443. eCollection 2021. PMID 34744918